CLINICAL TRIAL: NCT02641184
Title: A Multicenter Prospective Observational Study to Evaluate the Novel Risk Factors and Clinical Outcomes of Acute Myocardial Infarction (AMI)
Brief Title: Evaluation of Novel Risk Factors and Clinical Outcomes of Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Yangzhou No.1 People's Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Huaian first people's hospital (Unknown)
Responsible Party: Principal Investigator, Xiao Ye, MD, Doctor, Zhejiang Provincial People's Hospital
Other Study IDs: ZJPPH01
Record Dates: First submitted 2015-12-14; First posted 2015-12-29 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Acute Myocardial Infarction
Keywords: Myocardial Infarction; Cardiovascular Diseases; Heart Diseases; Infarction; Diabetes
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Cardiovascular Diseases; Heart Diseases; Infarction; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens for biomarker analysis and storage for future genetic studies
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate the potential novel risk factors for acute myocardial infarction. Predictors of poor outcomes will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Less than 12 hours after the onset of myocardial infarction symptoms
* Myocardial necrosis, as evidenced by increased Creatine Kinase Isoenzyme (CK-MB) or troponin levels

Exclusion Criteria:

* Age under 18 years-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to an emergency room and diagnosed as acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | maximum 5 years
  Composite of angina pectoris, reinfarction, unplanned rehospitalization, stent thrombosis, incidence of cardiac death in the duration of follow-up

SECONDARY OUTCOMES:
Length of hospital stay | in the phase of hospital stay, maximum 30 days
  The length of in-hospital stay is counted as a secondary outcome
New-onset diabetes | the duration of follow-up, maximum 5 years
  New-onset diabetes are defined as newly-diagnosed type 2 diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Baiming Qu, MD, Principal Investigator — Department of Cardiology, Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang provincial people's hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share data